CLINICAL TRIAL: NCT06359171
Title: Effectiveness of the ARTHE-e App for Exercise Adherence in People With Knee Osteoarthritis: Protocol for a Randomized Controlled Trial (ARTHe 3)
Brief Title: Effectiveness of the ARTH-e Application for Exercise Adherence in People With Knee Osteoarthritis : RCT
Acronym: ARTH-e3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RBHP 2023 LANHERS
Record Dates: First submitted 2024-02-13; First posted 2024-04-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; e-health; app; effectiveness
MeSH Terms: conditions — Osteoarthritis, Knee; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a multicenter, prospective, comparative, randomised trial (1:1). Participants will be randomized to one of two groups: control or experimental. In each group (control or experimental), each participant will be able to use the application for a period of 6 months.
  * Control group: physician's advice with examples of self-exercise (knee osteoarthritis booklet) + prescription for 12 physiotherapy sessions + delivery of a GARMIN connected bracelet.
  * Intervention group: download the application + adapted physical activity session with an APA/physiotherapist + delivery of the knee osteoarthritis booklet + prescription for 12 physiotherapy sessions + delivery of a GARMIN connected bracelet.
Who Masked: Investigator
Masking Description: The investigating physician who will carry out the inclusion visit will know the result of the randomization which will be carried out during the consultation. The second evaluator, who will carry out the end-of-study visit, will not know the patient's group. As a result, the assessment will be neutral and the second assessor will evaluate the patient without being influenced by the study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard care
- Experimental group (Experimental): Standard care and participants use the ARTH-e application for 6 months
  Interventions: Other: Application ARTH-e

INTERVENTIONS:
Other: Application ARTH-e — The ARTH-e application must be downloaded via the PlayStore or Applestore platform on phone and/or tablet. Once the application has been downloaded, the patient must scan a QRcode sent by the CHU to anonymize the data.
  Participants will have 6 months to use the application at their convenience.
  Arms: Experimental group

SUMMARY:
The aim of this study is to investigate the effectiveness of a smartphone-based e-health application (intervention group) compared with standard care (control group) in terms of changes in adherence in patients with knee osteoarthritis using the EARS questionnaire. In addition, other questionnaires presented in the appendix (KOOS, TSK, EPAP, EQ-5D-3L, pain) will be given to all patients in order to meet the secondary evaluation criteria.

DETAILED DESCRIPTION:
Knee osteoarthritis is the most common joint disease affecting the joint itself as well as the peri-articular structures in a global and progressive manner. It can affect all the joints of the body, with a predominance for those which undergo strong mechanical constraints such as the rachis, the hip or the knee. It is a chronic pathology correlated with age, since nearly one adult in two is affected by osteoarthritis.

Today, connected objects have taken a predominant place in the daily life of the majority of the population, including seniors. It is an object of communication and socialization as well as a major information tool. E-health applications are more and more numerous in the stores and are a tool for assistance, information and support already used in many fields. In the context of therapeutic education, it is a motivational tool that can accompany patients by adapting to their needs and progress compared to traditional self-exercise methods. Studies of the obstacles and levers for the use of smartphone applications in chronic pathologies such as low back pain support the development of this tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 40 and 85 years with uni or bilateral knee osteoarthritis according to EULAR (European League Against Rheumatism) criteria, symptomatic and diagnosed prior to inclusion by a specialist or not.
* Having an involvement of at least one knee.
* Own a smartphone or tablet running at least Android 5 or iOS 11.
* Able to give written consent to participate in the study.
* Beneficiary of a social security plan.

Exclusion Criteria:

* pregnant or breast-feeding women Patients under legal protection measures (guardianship, curatorship or protection of the court)
* Patients who have undergone knee surgery (total or partial prosthesis, tibial transposition surgery, arthrodesis)
* Patients with inflammatory rheumatism
* Patients with neurological sequelae
* Contraindications to physical activity for medical reasons
* Patients with difficulties in understanding the French language
* Refusal to participate
* Patients who have already participated in the ARTH-e 2 study or who are already included in a research protocol that could influence the current protocol

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Exercise Adherence Rating Scale | 6 months
  This questionnaire, validated in French, comprises 6 items. Scoring is based on a 5-point Likert scale (from 0 - "completely agree" to 4 - "completely disagree"). This results in a score ranging from 0 to 24. A higher score indicates greater support.
  The evolution of the score (i.e. the kinetics) will be compared between randomisation groups using a mixed model, taking into account the group, time and time x group interaction effects; it is therefore the value of EARS and not a variation that will be considered for the analysis.

SECONDARY OUTCOMES:
Exercise Adherence Rating Scale | 2 months and 4 months
  This questionnaire, validated in French, comprises 6 items. Scoring is based on a 5-point Likert scale (from 0 - "completely agree" to 4 - "completely disagree"). This results in a score ranging from 0 to 24. A higher score indicates greater support. The evolution of the score (i.e. the kinetics) will be compared between randomisation groups using a mixed model, taking into account the group, time and time x group interaction effects; it is therefore the value of EARS and not a variation that will be considered for the analysis.
EPAP questionnaire | Inclusion and 6 months
  Identification of barriers and levers to regular physical activity using the EPAP questionnaire. This questionnaire contains 24 items on the facilities and obstacles encountered when engaging in physical activity. The maximum score for this questionnaire is 100 points. Responses range from "Strongly disagree" (0 points) to "Strongly agree" (4 points). Responses to this questionnaire will be collected at inclusion and at the end of the study.
TSK questionnaire | Inclusion and at 6 months
  Evaluation of fears and anxieties related to pain that may be experienced during physical exercise using the TSK questionnaire at inclusion and at the end of the study. This questionnaire contains 17 statements. Patients were asked to circle the number that best corresponded to them (4 points). Responses ranged from "Strongly disagree" (1 point) to "Strongly agree" (4 points). The maximum score is 68. The higher the score, the greater the level of kinesiophobia.
Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire | Inclusion and 6 months
  Comparison of the functional evaluation collected at inclusion and at 6 months of use of the application via the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire. This questionnaire consists of 17 statements answering the question "Over the last eight days, how difficult́ have you beeń doing each of the following activities?". Responses range from "absent" (0 points) to "extreme" (4 points). The maximum score is 68. A high score is predictive of functional deterioration.
EQ-5D-3L questionnaire | Inclusion and at 6 months
  Evaluation of quality of life using the EQ-5D-3L questionnaire. This questionnaire consists of two aspects: a descriptive system (EQ-5D) and a visual analogue scale (EQ-VAS). The questionnaire comprises five dimensions: mobility, personal care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, a few problems and extreme problems. The patient therefore ticks the box that seems most appropriate to their current state.
Mobility | Inclusion and at 6 months
  Measurement of joint mobility with a goniometer (flexion/extension)
Average number of steps per day | Inclusion, 2,4,6 months
  Collection of average number of steps per day for 6 months during telephone calls (every 2 months). The GARMIN connected bracelet will allow us to collect the number of average steps per day (four measurement times over one week before each evaluation: inclusion, 2 months, 4 months and 6 months) via its GARMIN connect application.
Parameters for use of the ARTHE application | 2,4,6 months
  Collection of parameters for use of the ARTHE application, if applicable (for the intervention group), the number of sessions carried out per week will be collected by extracting data from the application's production back office.
Functional tests - 30 sec chair lifts | Inclusion and 6 months
  Functional tests: number of 30-second chair lifts at inclusion and at 6 months.The patient should remain in the sit-to-stand position for as long as possible (30 sec). The evaluator counts the number of sit-ups performed.
Functional tests - Stair Climbing Test | Inclusion and 6 months
  Functional tests: Stair Climbing Test (in seconds) at inclusion and at 6 months. The patient will be asked to climb 1The patient will be asked to climb 11 steps (height 13.5cm), make a U-turn and descend them as quickly as possible, while maintaining safety during the test (no loss of balance). Climbing and descending time will be measured separately with a stopwatch. 1 steps (height 13.5cm), make a half-turn and descend them as quickly as possible, but keeping safe during the test (without loss of balance). Climbing and descending times will be measured separately with a stopwatch.
Functional tests - 6MWT | Inclusion and 6 months
  Functional tests: 6-minute walk test (6 MWT) (in meters) at inclusion and at 6 months.This test carried out in a corridor with pads numbered from 1 to 60. The patient must walk back and forth for 6 minutes. The examiner measures the distance covered during these 6 minutes.
Functional tests - quadriceps isometric strength test with dynamometer | Inclusion and 6 months
  Functional tests: quadriceps isometric strength test (in N/Kg)with a dynamometer at inclusion and at 6 months. The participant will be asked to push the leg forward as hard as possible (isometric contraction of the quadriceps) for 5 seconds. Three trial contractions will be performed with progressive effort (weak, medium and strong). Then, three consecutive maximum contractions will be recorded using a dynamometer. The maximum value will be recorded and normalized in relation to the patient's body mass [N/kg].
Medico-economic analysis | Inclusion and 6 months
  Medico-economic analysis carried out using a data record (drug management, medical consultations, hospitalisations, use of alternative therapies, additional examinations, use of medical transport).
Pain Visual Analog Scale | Inclusion, 2 months, 4 months and 6 months
  Change in the average level of pain over the last 3 days collected during the telephone interview using a 10-point Numerical Scale (0 = "No pain" to 10 = "Maximum imaginable pain") at inclusion, 2 months, 4 months and 6 months of use of the application.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Emile Roux, Le Puy-en-Velay
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelletier-Visa M, Dobija L, Bonhomme A, Lanhers C, Pereira B, Coudeyre E. Effectiveness of the ARTHE-e app for exercise adherence in people with knee osteoarthritis: protocol for a randomised controlled trial. BMJ Open. 2025 Jan 20;15(1):e088860. doi: 10.1136/bmjopen-2024-088860. PMID 39832974